CLINICAL TRIAL: NCT03248258
Title: Enhancing Shared Decision-Making in Metastatic Breast Cancer (Qualitative Study)
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Gabrielle Rocque, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-170518009
Record Dates: First submitted 2017-07-26; First posted 2017-08-14 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Decision Making ,Shared; De-escalation
Keywords: Metastatic Breast Cancer; Treatment Decision Making; Shared Decision Making; Early Stage Breast Cancer; De-escalation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Metastatic Breast Interview Participants - Shared Decision Making: Metastatic Breast Patient Participants will be interviewed on the topic of Shared Decision Making. This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Early Stage Breast Interview Participants - Shared Decision Making: Early Stage Breast Patient Participants will be interviewed on the topic of Shared Decision Making. This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Provider Focus Group -Shared Decision Making: Clinic Provider Participants will participate in a focus group on the topic of Shared Decision Making. This will be a one time, focus group interview with a trained moderator.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Non-UAB Provider Shared Decision Making: Non-UAB Provider Participants will be interviewed on the topic of Shared Decision Making. This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Early Stage de-escalation Interview Participants: Early Stage Breast Patient Participants will be interviewed on the topic of de-escalation of cancer treatment. This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Patient Advocate de-escalation Interview Participants: Patient Advocate Participants will be interviewed on the topic of de-escalation of cancer treatment. This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Physician de-escalation Interview Participants: Physician Participants will be interviewed on the topic of de-escalation of cancer treatment. This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions
- Early Stage Feedback Interview Participants: Early Stage Breast Patient Participants will be interviewed to provide feedback on a decision making tool (video). This will be a one time, one-on-one interview with a trained interviewer.
  Interventions: Other: Qualitative Interview or Focus group discussions

INTERVENTIONS:
Other: Qualitative Interview or Focus group discussions — The purpose of this study is to identify factors that influence decision-making in treatment selection and the optimal approach for sharing information about prognosis and guideline-based care.
  Secondly, to further understand patient perspective on the concept of de-escalation, in which patients reduce the amount of chemotherapy to avoid side effects and (2) consider how prognosis would impact their decision-making about reducing chemotherapy (as standard or care or within a clinical trial).

SUMMARY:
Develop a Metastatic Breast Cancer (MBC)-specific electronic Treatment Plans (TP).

Phase 1:

Aim 1a: Patient interviews along with navigator, nurse, and physician focus group discussions will be used to identify factors that influence decision-making in treatment selection and the optimal approach for sharing information about prognosis and guideline-based care. Identify decisional needs for Shared Decision Making (SDM) in MBC. Investigators will conduct semi-structured interviews/discussion groups with patients, navigators, nurses, and physicians to elements important to decision-making.

Phase 2:

Aim 1b: Develop MBC-specific TP. Investigators will build upon Aim1a to systematically develop the TP intervention using the Ottawa Decision Support Framework. Investigators will test the TPs with 5 patients and conduct qualitative investigations to refine the TP using an iterative process.

Phase 3:Further explore decision-making related to reducing amount of chemotherapy for patients with good prognosis.

DETAILED DESCRIPTION:
Phase 1:

Investigators will use patient interviews and navigator, nurse, and physician focus group discussions to identify factors that influence decision-making in treatment selection and the optimal approach for sharing information about prognosis and guideline-based care. Patients will be recruited from the medical oncology clinic. Patients will be identified by their primary oncologist. All eligible patient will be provided with a study information flyer. All patient participants will be asked to provide written informed consent prior to participation in interviews; provider participants will be provided with Information sheets prior to focus groups by a research coordinator. Participants in Group 1 will be asked to complete a demographic form. The demographic forms for patients, navigators, nurses, and medical oncologists are included in Appendix B. Demographic form will include questions about your age, sex, race and education. The demographic form will take 5 minutes to complete. At study entry, descriptive data including patient demographics (age, sex, race), breast cancer characteristics (subtype, line of therapy, specific treatment offered, prior treatments received), physician will be collected to provide clinical context for the analysis. The patients will be interviewed at the patient's next appointment (either with the physician or in the infusion center) or the patients can schedule to come on an off clinic day of their preference. The study coordinators will offer each patient the option to complete the consent form at home. If they decide to complete the consent form at home investigators will follow up with by contacting them on the telephone to ensure that the consent form was completed and to confirm their interview at their next clinic visit or an off day of their preference. This 30 minute to an hour interview will take place in a private meeting room within the UAB Comprehensive cancer center. The patient interviews will be audio-recorded by using a digital audio recorder.

Phase 2:

Patients will be recruited from the medical oncology clinic. Patients will be identified by their primary oncologist. A trained research coordinator will consent the patient during a routine clinic visit. This group will consist of 5 new patients who did not participate in Group 1 patient interviews. Descriptive data including patient name and medical record number will be collected on a tracking sheet. No other personal identifiable information will be collected. This 30-minute interview will take place in the clinic room or a private room within the UAB Comprehensive cancer center (based on patient preference). The researcher will provide the patient with the iPad for completion of baseline patient-reported outcome questionnaires using the Carevive® platform for a test patient in a test environment which will not be linked to the patient's medical record. The intervention questionnaire will include standard questions used to routine treatment planning at UAB/MCI as well as any study-specific questions generated from Phase I above. This will allow feedback on the questionnaire itself. The research coordinator will then provide the patient with an example TP that includes responses to the questionnaire. The study PI will review the electronic or a printed version with the patient to get feedback on the acceptability of the TP, content of the TP, and the best approach to utilizing the TP. This process may be modified based on results of our qualitative analysis.

Investigators will conduct separate focus groups with each provider group. This will include 7 breast medical oncologists, 10 patient navigators, and 10 nurses (5 clinic nurses who work directly with the breast oncologists and 5 infusion nurses).

Phase 3:

The purpose of this phase is to (1) further understand patient perspective on the concept of de-escalation, in which patients reduce the amount of chemotherapy to avoid side effects and (2) consider how prognosis would impact their decision-making about reducing chemotherapy (as standard or care or within a clinical trial). This study will include both patients and patient advocates, who bring a broad perspective to how the patient experience should be considered in research. Interviews with patients, patient advocates, and physicians will be conducted either in person or by phone/zoom based on patient preference. In person patient interviews will be conducted (1) in the UAB Medical Oncology outpatient clinic rooms or in private room in the UAB Comprehensive Cancer Center (based on patient preference for location). In person patient advocate or physician interviews will be conducted at in-person meetings of the Eastern Cooperative Group, which are routinely attended by the patient advocates and physicians in the private room or location of the advocate's choice.

ELIGIBILITY:
Patient Criteria (Phase I,II,III):

Inclusion Criteria:

* 1. Women with age ≥ 18
* 2. Presence of Metastatic Breast Cancer or Early Stage Breast Cancer
* 3. Patients may be receiving any line and type of therapy including both standard of care and clinical trials.

Exclusion Criteria:

* 1. Patient who are not able to read and/or speak English
* 2. Patients with a life expectancy less than 3 months
* 3. Patients unable to provide informed consent
* 4. Men

Patient Advocates (Phase III)

Inclusion criteria:

1. Providers who are self-identified patient advocates working with breast cancer researchers

Exclusion criteria:

1. None

   Sampling: We will conduct interviews with 10-20 patient advocates for phase 3 of this project.

   Provider (navigator, nurse, physician) (Pjhase I, III)

   Inclusion criteria:
2. Providers who have direct contact with breast cancer patients

Exclusion criteria:

2. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient Participant Groups are women only
Study Population: Metastatic and Early stage Breast Cancer patients receiving care at UAB Hematology/Oncology Kirklin Clinic. Breast Cancer Patient advocates, oncology nurses, navigators, and Oncology Physicians
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Shared Decision Making | 3 years
  Shared decision making occurs when patients are informed of risks and benefits associated with treatment options and partner with their oncologist to incorporate their personal preferences and values into decision-making. Shared decision making in medicine can improve quality of care and reduce costs. This will be accessed using qualitative interviews and focus groups discussions. This is not a survey based study.
Concept of de-escalation | 2 years
  Patients reduce the amount of chemotherapy to avoid side effects

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle B Rocque, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rocque GB, Andrews C, Lawhon VM, Ingram SA, Frazier RM, Smith ML, Wagner LI, Zubkoff L, Wallner LP, Wolff AC. Physician Perspectives on Reducing Curative Cancer Treatment Intensity for Populations Underrepresented in Clinical Trials. Oncologist. 2022 Dec 9;27(12):1067-1073. doi: 10.1093/oncolo/oyac191. PMID 36215065